CLINICAL TRIAL: NCT02862119
Title: Ffr-gUidance for compLete Non-cuLprit REVASCularization - a Registry-based Randomized Clinical Trial
Brief Title: Ffr-gUidance for compLete Non-cuLprit REVASCularization
Acronym: FULL REVASC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Felix Bohm (Other)
Collaborators: Uppsala University (Other); The Swedish Research Council (Other Government); Swedish Heart Lung Foundation (Other); Abbott (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Felix Bohm, MD, PhD, Interventional Cardiologist, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FULL REVASC
Record Dates: First submitted 2016-08-01; First posted 2016-08-10 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Coronary Artery Disease; ST-elevation Myocardial Infarction
Keywords: percutaneous coronary intervention; fractional flow reserve; all cause mortality; myocardial infarction; registry-based randomized clinical trial
MeSH Terms: conditions — Coronary Artery Disease; ST Elevation Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR Treatment Arm (Experimental): Following PCI of the infarct related artery it is up to the PCI operator to perform FFR-guided PCI of non-infarct related lesion(s) during the index procedure or later during the index hospital admission. For stenosis grade 90-99% FFR is not mandatory (but recommended). An FFR value of ≤0.80 is to be considered significant for ischemia with a recommendation that non-culprit PCI is performed. It is up to the operator to decide whether to use intra-venous or intracoronary adenosine during FFR. An FFR of >0.80 is to be considered non-significant for ischemia with a recommendation that medical management is pursued.
  Pressure wires: Only Fractional Flow Reserve pressure wires from St Jude Medical or Boston Scientific can be used in this study.
  Interventions: Procedure: FFR Treatment Arm
- Conservative Treatment Arm (Active Comparator): Only the infarct-related artery will be treated with PCI in this treatment arm during the index hospital admission. Medical therapy for angina pectoris is at the investigators discretion. Clinical follow-up of symptoms is recommended, but it is also acceptable to make a plan at hospital discharge for a later outpatient non-invasive stress-test. It is not acceptable to plan for an elective PCI in this treatment arm without signs of ischemia or symptoms.
  Interventions: Other: Conservative Treatment Arm

INTERVENTIONS:
Procedure: FFR Treatment Arm — Fractional Flow Reserve-guided PCI of non-culprit lesions during index hospital admission
  Arms: FFR Treatment Arm
Other: Conservative Treatment Arm — Initial Conservative management of non-culprit lesions during index hospital admission
  Arms: Conservative Treatment Arm

SUMMARY:
Background: The best strategy for ST-elevation myocardial infarction (STEMI) patients with multi-vessel disease, who undergo primary percutaneous coronary intervention (PCI) of the infarct-related artery (IRA) in the acute phase with remaining multivessel disease, is still not well established. Current guidelines recommend PCI of only the infarct related artery (IRA). However, recent small scale randomised controlled trials indicate that full revascularization of these non-infarct related arteries during the index procedure is superior to initial conservative treatment. Fractional flow reserve (FFR), a method used to determine ischemia-inducing lesions, has been shown to be superior to angiography-guided PCI in stable angina.

Objective and methods: To test the hypothesis that a strategy of systematic complete revascularization with FFR-guided PCI following STEMI/very high risk NSTEMI leads to improved clinical outcomes compared to initial conservative management of non-culprit lesions. The trial is a prospective international multicentre registry-based randomized controlled trial with combined primary endpoint of all-cause mortality, or non-fatal MI, or unplanned revascularization at a minimum follow-up of 2-3 years. The first key secondary endpoint is the combined endpoint of all-cause mortality or myocardial infarction. The second key secondary endpoint is unplanned revascularization. 1542 patients with acute STEMI/very high risk NSTEMI with multi-vessel disease in Sweden, Denmark, Serbia, Finland, Latvia, Australia and New Zealand will be randomized into 2 arms:

1. FFR-guided PCI of non-culprit lesions during index hospital admission or
2. Initial conservative management following acute PCI of the culprit lesion(s) or

Randomization and data collection in the registries - the Swedish Coronary Angiography and Angioplasty Registry (SCAAR) and corresponding registries in other countries (or electronic data capture) - will ensure low bias, high inclusion rate and excellent follow-up of events at a low cost. Adjudication of clinical events and collection of data from other registries including death cause registries is also planned.

Significance: If this study shows that FFR-guided PCI of non-culprit lesions in STEMI/very high risk NSTEMI improves clinical outcome compared to conventional management this will change practise in how we should best manage these patients. Therefore a study of this size will definitely be of great importance in determining future guidelines for this large patient group to reduce both morbidity and mortality.

DETAILED DESCRIPTION:
Background Information: Early epicardial coronary reperfusion is a prerequisite for the effective salvage of ischemic myocardium and reduces morbidity and mortality in patients with ST elevation myocardial infarction (STEMI). The recent ESC guidelines currently recommend percutaneous coronary intervention (PCI) of only the infarct related artery (IRA) in the setting of acute ST-elevation myocardial infarction (STEMI). Subsequent management of residual disease is initially conservative with a low threshold for non-invasive investigation for residual ischemia. There is a recent meta-analysis of 34279 patients with 1819 cardiovascular deaths registered during follow-up showing that PCI of the culprit lesion only is associated with reduced mortality as compared to full revascularization at the time of STEMI in multivessel disease. Also in non ST-segment elevation myocardial infarction (NSTEMI), the strategy of multivessel PCI for suitable significant stenoses-rather than PCI limited to the culprit lesion-has not been evaluated in an appropriate, randomized fashion according to the European Society of Cardiology guidelines on myocardial revascularization. In NSTEMI there is growing evidence to suggest a benefit of an invasive strategy within 2 h in patients with a very high risk profile according to the ESC NSTEMI guidelines. Accordingly, also patients with a very high risk NSTEMI requiring urgent revascularization may be included in the current study.

Recent small scale randomised controlled trials (RCT) have however produced results which suggest that in cases where there is anatomically significant non-culprit multi-vessel disease full revascularization of these non-infarct related arteries during the index procedure or at least during the same hospitalization is superior to initial conservative treatment. Since these studies were so small and also go against earlier observational studies and current guidelines it is therefore difficult to draw any conclusions on how to treat this patient group in the optimal way to reduce mortality.

By way of paradox, in recent years it has been shown that fractional flow reserve (FFR) used to determine ischemia-inducing lesions is superior to angiography guided PCI in both stable angina and in NSTEMI. Whether performing full revascularization of physiologically significant non-culprit lesions for patients with STEMI improves outcome compared to an initial conservative approach is not known. The primary PCI in multivessel disease study(PRIMULTI) was a small study (650 patients) that investigated this question with a combined primary endpoint of all cause death, myocardial infarction or revascularization at one year. In PRIMULTI conservative treatment was safe; there was no difference at all regarding death and myocardial infarction, only revascularization. One critique of these studies is that they are including revascularization in the primary endpoint and it is expected that you will increase revascularization if you leave significant stenoses untreated. The key question is if complete revascularization prevents death or MI.

Therefore, the aim of this study is to investigate whether in patients with STEMI/rescue PCI/risk evaluation following successful thrombolysis/very high risk NSTEMI FFR-guided PCI of non-culprit lesions during the index hospital admission will improve cardiovascular outcomes compared to an initially conservative approach of non-culprit lesions. The study aim is powered statistically for the combined primary endpoint of total mortality and myocardial infarction (MI) at a minimum follow-up of 1 year (all events when the last patient has been for 1 year).

Assessments and Procedures:

All patients will undergo primary PCI according to clinical routine for patients with STEMI/Rescue PCI/Risk evaluation following successful thrombolysis/very high risk NSTEMI. If index procedure PCI is performed then oral informed consent of the study will be obtained and the patient will be randomized following PCI of the culprit lesion.

A simple randomization procedure based on a computer module will be performed via SCAAR registry (Sweden). Other participating countries without possibility to randomize patients through registries can do this through a web page. It is strongly recommended that randomization is done directly following primary PCI of the culprit lesion. However, it is possible to randomize the patient within 6 h from puncture time of the index procedure.

The patients will receive written information about the study and sign a consent form in the ward after the PCI procedure is performed.

Follow-up of both treatment arms: If patients at follow-up are found to have angina pectoris that could not be medically managed, it is recommended that an imaging-based non-invasive stress test is performed before deciding on a new elective coronary angiography according to current guidelines. If patients in both groups are found to have signs of significant ischemia on a stress-test or still have significant angina and sent for elective coronary angiography, then FFR is allowed according to current ESC guidelines of stable coronary artery disease and is at the discretion of the patient responsible physician. However, it is recommended that a non-invasive stress test is performed as first option if a patient comes back with angina.

Patients who are eligible but not randomized into the study will be followed in the registries for the same endpoints.

Data will be collected for all patients on hospitalization for myocardial infarction from the The Swedish Web-system for Enhancement and Development of Evidence- based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART) registry (Sweden) or corresponding registries in other countries.

Data will also be collected from the the Swedish Coronary Angiography and Angioplasty Registry (SCAAR) in Sweden or corresponding registries in other countries.

Data on coronary-artery bypass surgery after the index procedure will be determined by the diagnose registry or CABG registry in Sweden. For deceased patients data on cause of death will be collected from the Swedish Death Cause Registry. Corresponding registries in other countries will also be used where possible.

Other participating countries must decide their possibility to capture registry data from corresponding registries according to the data model for the study. If not possible data must be collected manually through an UCR EDC system that mirrors the interface in registries used in Sweden.

Treatment assignment:

Randomization (1:1) will be performed by means of an online randomization module within the SCAAR registry using permuted block randomization stratified by site. In other participating countries randomization will be performed in corresponding registries or through a web page.

Intention-to-treat analysis will be performed as primary analysis.

A research nurse at each site will contact each patient and perform a medical record review at 30 days and one year to confirm if the patient has experienced anything of the following:

MI, unplanned rehospitalization due to anything of the following: revascularization, major bleeding requiring transfusion or surgery, stroke or heart failure. Furthermore, the Seattle Angina Questionnaire-7 will be used to evaluate effects on angina pectoris.

A majority of patients aged <75 years in the study will have a clinical follow-up visit at one year to a Cardiology nurse. This is according to clinical routine for patients in Sweden with and age <75 years. At this visit quality of life parameters (EQ-5D) will be entered into the the Swedish quality registry for secondary prevention according to clinical routine.

The data safety monitoring board (DSMB) will have the possibility to stop enrolment due to perceived increased risk to patients in the FFR-group only.

No follow-up of adverse events is planned.

All MIs and unplanned revascularization (PCI/CABG) will be adjudicated by the Clinical Events Adjudication (CEA) group at Uppsala Clinical Research Centre (UCR). The CEA charter defines the specific criteria and definitions of the endpoints. The adjudication decision will be entered in a CEA database, handled by UCR. All details of the event definitions and the adjudication process are described in detail in the CEA charter.

Data management:

Data defined as study data will be recorded in an electronic data capture system (EDC) at UCR. Access to data sets with information on allocated treatment, or data summaries presented by treatment, will be restricted and documented to decrease the risk of bias due to non-blinded decisions during the study.

Data will be evaluated for compliance with the protocol and accuracy in relation to source documents which means that regular data checks for completeness of the variables in the EDC system will be done and follow-up of informed consent. The study will be conducted in accordance with procedures identified in the protocol. Regular monitoring will be performed. Following written standard operating procedures, the monitors will verify that the clinical trial is conducted and data are generated, documented and reported in compliance with the protocol and the applicable regulatory requirements.

Statistical analyses:

Analyses will primarily be performed on the intention-to-treat (ITT) set, defined as all intentionally randomized patients, by randomized treatment. All statistical tests will be performed on the 5% significance level using two-sided tests.

All endpoints will be presented as Kaplan-Meier plots and frequency tables at 30 days and 1 year, by randomized treatment, and analysed using Cox proportional hazards regression with randomized treatment, country, and gender as factors, and age as a continuous covariate, and treatment contrasts presented as hazard ratios with 95% confidence interval and associated p-values. The primary analysis will be based on events of all follow-up time of each patient at time of data base lock.

The sample size calculation is based on the patients with 2- or 3-vessel disease in the TASTE trial. This group constitutes 3138 patients, of which 208 died and 312 had a composite event of death or rehospitalization with myocardial infarction within 1 year.

4052 patients (2026 per arm) would give 80% power to detect a relative risk reduction of 25% at one year in the composite of all-cause death and myocardial infarction, for FFR-guided non-culprit PCI against conservative treatment.

Following publication of the COMPLETE trial in September 2019, enrollment into the FULL REVASC trial was stopped. See publication in American Heart Journal 2021 - FULL REVASC Design and Rationale, Böhm et al. for details. A new power calculation was performed and the 1,542 patients will be followed for at least 2.75 years after last patient in (june 2022) to reach at least a total of 346 events (death, MI and unplanned revascularization). The study is now event driven and the combined primary endpoint is changed to also include unplanned revascularization.

Before starting the study all centres will have a web-based start meeting with presentation of the study, study procedures and documentation (Investigator Study File with Essential Documents). The sponsor is responsible for performing remote monitoring, no on-site monitoring is planned. Data from the randomization module (registry data) will be evaluated for protocol compliance and logs for signed informed consents will be sent to Sponsor for follow-up. The monitoring activities will be described in detail in the monitoring plan.

The Investigator or designee (PCI operators) will record data from the source into the SCAAR registry or through an EDC system in countries outside the SCAAR platform. Data fields should not be left blank. Also, discharging doctors will record data in the Swedish Register of Information and Knowledge about Swedish Heart Intensive Care Admissions and in corresponding registries in other participating countries. Data will be entered in Heart Surgery Registries for patients with CABG (in Sweden and in other countries where possible).

The statistician will analyse the original registry data regarding components of the primary endpoint and report to the DSMB.

ELIGIBILITY:
Inclusion Criteria:

The following specific criteria must be fulfilled:

1. Symptoms indicating acute myocardial ischemia with a duration >30 min and occurring ≤ 24 h prior to randomization or presentation.
2. One of the following:

   1. STEMI: ST elevation above the J-point of ≥0.1 millivolt in ≥ two contiguous leads or left bundle branch block
   2. Rescue PCI
   3. Risk evaluation following successful thrombolysis
   4. Very high risk NSTEMI: dynamic ECG changes or ongoing chest pain or acute heart failure or hemodynamic instability independent of ECG changes or life-threatening ventricular arrhythmias.
3. PCI performed of infarct-related artery.
4. One or more non-culprit lesions at least 2.5 mm on angiogram (visually assessed as 50-99%) amenable for PCI.
5. Age >18 years.
6. Ability to provide informed consent.

Exclusion Criteria:

1. Previous CABG.
2. Left main disease of >50% stenosis requiring intervention.
3. Cardiogenic shock necessitating therapy in addition to revascularization. (LV support device or vasopressors).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1542 (Actual)
Dates: Start 2016-08-08 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Combined endpoint of all-cause mortality, or myocardial infarction, or unplanned revascularization. | Minimum 2-3 years
  Combined endpoint of all-cause mortality, or myocardial infarction, or unplanned revascularization during a minimum follow-up of 2-3 years.

SECONDARY OUTCOMES:
Combined endpoint of all-cause mortality, or myocardial infarction. | Minimum 2-3 years.
  Key Secondary Endpoint is Combined endpoint of all-cause mortality, or myocardial infarction. during follow-up. All suspected myocardial infarctions will be adjudicated.
Number of patients with unplanned revascularization (PCI/CABG) of the coronary arteries | Minimum 2-3 years.
  Key Secondary Endpoint is unplanned revascularization (PCI/CABG) during follow-up. All unplanned revascularizations will be adjudicated.
Combined end point of all-cause mortality, MI, and unplanned revascularization (PCI/CABG) at a minimum follow-up of 2-3 years in pre-specified subgroups | Minimum 2-3 years.
  Other Secondary Endpoint.
All-cause mortality | Minimum 2-3 years.
  Other Secondary Endpoint.
Myocardial infarction (fatal and non-fatal) | Minimum 2-3 years.
  Other Secondary Endpoint.
Cardiovascular mortality | Minimum 2-3 years.
  Other Secondary Endpoint.
Any revascularization (PCI/CABG) | Minimum 2-3 years.
  Other Secondary Endpoint.
Stent thrombosis (all treated vessels including nonculprit vessels) | Minimum 2-3 years.
  Other Secondary Endpoint.
Instent restenosis (all treated vessels including nonculprit vessels) | Minimum 2-3 years.
  Other Secondary Endpoint.
Target vessel revascularization (all treated vessels including nonculprit vessels) | Minimum 2-3 years.
  Other Secondary Endpoint.
Rehospitalization due to heart failure | Minimum 2-3 years.
  Other Secondary Endpoint.
Angina pectoris according the Seattle Angina Questionnaire-7 (SAQ-7) | Minimum 2-3 years.
  Other Secondary Endpoint.
Length of index hospital stay | 1 month
  Other Secondary Endpoint.
Quality of life according to the questionnaire EQ-5D at nurse visit at two months and/or one year for those patients that are registered in SEPHIA (Sweden only). | Minimum 2-3 years.
  Other Secondary Endpoint. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Health Economic evaluation of direct and indirect costs during follow-up | Minimum 2-3 years.
  Other Secondary Endpoint. The direct costs refer to those costs incurred as a result of medical management of the disease, drugs, admissions, complementary tests, patient transportation. Indirect costs refer to resources that are indirectly lost as a result of the disease or treatment, such as impaired ability to work or loss of production, in cases where people are unable to work due to the disease or the treatment.

OTHER OUTCOMES:
Contrast volume | 1 month
  Safety Outcome during index hospitalization
X-ray duration | 1 month
  Safety Outcome during index hospitalization
Neurological complications | 1 month
  Safety Outcome during index hospitalization
New renal insufficiency during index hospitalization | 1 month
  Safety Outcome during index hospitalization
Major bleeding (fatal, intracranial, or requiring operation/transfusion) | Minimum 2-3 years.
  Safety Outcome during entire follow-up
Stroke | Minimum 2-3 years.
  Safety Outcome during entire follow-up
Rehospitalization due to heart failure | Minimum 2-3 years.
  Safety Outcome during entire follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Felix Bohm, MD, PhD, Principal Investigator — Karolinska Institutet; Stefan James, Professor, Study Chair — Uppsala University, Sweden; Andreas Rück, MD, PhD, Study Director — Karolinska University Hospital; Thomas Engstrøm, MD, PhD, Study Director — Rigshospitalet, Denmark; Mika Laine, MD, PhD, Study Director — Helsinki University Hospital, Finland; Andrejs Erglis, Professor, Study Director — Riga, Latvia; Goran Stankovic, Professor, Study Director — Belgrade, Serbia; Carl Schultz, Professor, Study Director — Perth, Australia; Madhav Menon, MD, PhD, Study Director — Hamilton, New Zealand
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be confidential. Only data on Group level will be presented in scientific publications.

REFERENCES:
- [Derived] Bohm F, Mogensen B, Engstrom T, Stankovic G, Srdanovic I, Lonborg J, Zwackman S, Hamid M, Kellerth T, Lauermann J, Kajander OA, Andersson J, Linder R, Angeras O, Renlund H, Erglis A, Menon M, Schultz C, Laine M, Held C, Ruck A, Ostlund O, James S; FULL REVASC Trial Investigators. FFR-Guided Complete or Culprit-Only PCI in Patients with Myocardial Infarction. N Engl J Med. 2024 Apr 25;390(16):1481-1492. doi: 10.1056/NEJMoa2314149. Epub 2024 Apr 8. PMID 38587995
- [Derived] Ong P, Martinez Pereyra V, Sechtem U, Bekeredjian R. Management of patients with ST-segment myocardial infarction and multivessel disease: what are the options in 2022? Coron Artery Dis. 2022 Sep 1;33(6):485-489. doi: 10.1097/MCA.0000000000001157. Epub 2022 Jul 11. PMID 35811565
- [Derived] Bohm F, Mogensen B, Ostlund O, Engstrom T, Fossum E, Stankovic G, Angeras O, Erglis A, Menon M, Schultz C, Berry C, Liebetrau C, Laine M, Held C, Ruck A, James SK. The Full Revasc (Ffr-gUidance for compLete non-cuLprit REVASCularization) Registry-based randomized clinical trial. Am Heart J. 2021 Nov;241:92-100. doi: 10.1016/j.ahj.2021.07.007. Epub 2021 Jul 24. PMID 34310907